CLINICAL TRIAL: NCT05404997
Title: Comparative Effects of Shockwave Therapy and Maitland's Lumbar Mobilization on Pain, Disability and Range of Motion in Patients With Mechanical Low Back Pain
Brief Title: Comparative Effects of SWT and Maitland LM in Mechanical LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0127
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Low Back Pain
Keywords: low back pain, lumbar mobilization, shockwave therapy
MeSH Terms: conditions — Low Back Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave Therapy (Experimental): Common Treatment : Conventional physical therapy (lumbar stretching exercises and core strengthening exercises) Group A: Shockwave Therapy
  Interventions: Device: Shockwave Therapy
- Maitland's Lumbar Mobilizations (Experimental): Common Treatment: Conventional Physical Therapy (lumbar stretching exercises and core strengthening exercises) Group B: Maitland's Lumbar mobilizations
  Interventions: Other: Maitland's lumbar mobilizations

INTERVENTIONS:
Device: Shockwave Therapy — Subjects in Group A will receive conventional physical therapy treatment that involves lumbar stretching exercises (bridges, knee to chest, press-up back extensions, bird dogs) and core strengthening exercises (partial crunches, pelvic tilts, wall sits, hip stretches) for ten minutes. After the conventional therapy, this group will be given shockwave therapy treatment twice a week for four weeks.
  After exposing and cleaning the treated area with alcohol, adequate amount of gel will be placed on the lower back region, and the machine will be adjusted at (2000 shock per session, 8 sessions 2 per week for 4 weeks, energy flux density 0,18mJ per mm square, 2 bars of pressure, frequency 10hz), with using 20mm D-Actor head.
  Arms: Shockwave Therapy
Other: Maitland's lumbar mobilizations — Subjects in Group B will receive conventional physical therapy treatment that involves lumbar stretching exercises (bridges, knee to chest, press-up back extensions, bird dogs) and core strengthening exercises (partial crunches, pelvic tilts, wall sits, hip stretches) for ten minutes.
  After the conventional treatment, Group B will be given Maitland's lumbar postero-anterior glide mobilizations initiating from Grade 1, with 3-4 sets of oscillations of 40 counts in each set, 2 sets of oscillations will be given below and above the affected joint level.This whole mobilization treatment will also be given twice a week for 10 minutes.
  Arms: Maitland's Lumbar Mobilizations

SUMMARY:
Low back pain is a common neuro-musculo-skeletal problem affecting 40% of world's population at some point in their life and causes significant disability with loss of productive working hours. Low back pain is usually non-specific or mechanical and its mechanical origin is identified by the presence or absence of signs and symptoms i-e local or radicular pain, tenderness, spasm associated with different postures or movements. This study aims to compare the therapeutic effects of shockwave therapy and Maitland lumbar mobilizations on pain, disability and range of motion in patients having mechanical low back pain.

Current study will be randomized clinical trial in which convenience sampling technique will be used. Sample size will be 26. Subjects with age group of 25 to 45 years and who meet the inclusion and exclusion criteria will be included in this study and they will be randomly allocated into two groups. Group A will be given shockwave therapy treatment, while the group B will be given Maitland lumbar PA glide mobilizations. Each groups will also receive the conventional physical therapy treatment that includes lumbar stretching exercises and core strengthening exercises. Both the therapeutic techniques will be conducted for 4 weeks, two sessions per week for each group. Before, after two weeks and after four weeks of the treatment sessions, effects of treatment will be noted and quantitative data will be analyzed using SPSS software version 25.

DETAILED DESCRIPTION:
Low back pain (LBP) is increasingly becoming one of the main health concerns nowadays. It affects daily life and work routine and leads to medical consultations. The prevalence of NSLBP is approximately 10 to 25% in young and middle-aged individuals. Even though degenerative changes are minimal in this age group, more physical activities consequently make this group vulnerable to various physical strains. Approximately 10% of LBP cases have an identifiable pathology, while the remaining 90% are non-specific LBP (NSLBP), reflecting LBP of unknown underlying pathology, characterized by pain, muscle tension, and stiffness between 12th rib and inferior gluteal fold. Based on duration, LBP can be categorized as acute (less than six weeks), sub-acute (six to twelve weeks), and chronic (more than twelve weeks). Common symptom is the pain that gets worse with activity and relieved by rest. There are different methods for LBP treatment like surgery, oral medication, injection at lumbar region, psychotherapy, chiropractic and physiotherapy. Physiotherapy modalities and techniques like electrotherapy, low level laser, ultrasound, massage, shortwave, traction, superficial heat, spinal manipulation and exercise therapy are used to treat such cases. Extracorporeal Shock Wave Therapy (ESWT) has emerged as a popular tool for treatment of musculoskeletal disorders such as lateral epicondylitis, painful shoulder syndrome and plantar fasciitis. The two primary types of shock waves are the Focused Extracorporeal Shock Wave (fESW) and the Radial Extracorporeal Shock Wave (rESW). They differ in terms of the manner and extent of the acoustic energy propagation, the shape of the beam and its physical properties. Maitland mobilization techniques are thought to benefit patients with lumbar mechanical pain through the stimulation of joint mechanoreceptors.

A systematic review and meta-analysis of RCTS was conducted in 2020 to check the effectiveness and safety of extracorporeal shockwave treatment on low back pain. Multiple electronic databases including PubMed, Embase, Cochrane's library, China National Knowledge Infrastructure (CNKI), and Wan Fang Data were searched until December, 2019 to identify studies assessing the effectiveness and safety of EPSW for LBP. The main outcome was pain intensity which was measured using visual analogue scale (VAS) and numeric pain rating scale (NPRS).Functional status, quality of life and psychological outcomes were also measured using oswestry disability index (ODI). Findings of all these studies concluded that the use of focused ESWT is effective in alleviating pain and improving general functional state of patients with low back pain. The effectiveness of Maitland spinal mobilization therapy in the treatment of non-specific low back pain. It was a prospective study that involved ninety (90) subjects who completed the recommended four-week program. All subjects were given spinal mobilization therapy using Maitland method. The conclusions of this study indicated that manual therapy is a consideration in treatment of non-specific LBP and as an alternative to conventional treatment methods.

The effects of shockwave therapy and Maitland lumbar mobilizations have been seen to be the effective approaches in the treatment of mechanical or non-specific low back pain. But these treatment approaches have seen independently in treating low back pain. But there is no literature available that compares the effect of both techniques. So to see the comparative effects of these two techniques will be the main goal of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-45 years
* Gender: both male and female
* Patients that reports in physiotherapy OPD or referred from orthopedic department, diagnosed with mechanical low back pain having pain for more than 2 weeks.

Exclusion Criteria:

* Patients with surgical interventions to lumbar vertebral region.
* Spondylosis
* Disc prolapse
* Spondylolisthesis
* Spinal tumor or inflammatory disease such as rheumatism

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 10 Months
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain". NPRS have shown high test-retest reliability (r = 0.96 and 0.95, respectively)
Oswestry Disability Index (ODI) | 10 Months
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools The final score/index ranges from 0-100.
  A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound
Bubble Inclinometer | 10 Months
  The simple bubble inclinometer has excellent clinical reliability (ICC >.90) for measuring lumbar lordosis and thoracic kyphosis in standing.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- Bin Inam's Clinic, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baig AAM, Ahmed SI, Ali SS, Rahmani A, Siddiqui F. Role of posterior-anterior vertebral mobilization versus thermotherapy in non specific lower back pain. Pak J Med Sci. 2018 Mar-Apr;34(2):435-439. doi: 10.12669/pjms.342.12402. PMID 29805422
- [Background] Bhat P V, Patel VD, Eapen C, Shenoy M, Milanese S. Myofascial release versus Mulligan sustained natural apophyseal glides' immediate and short-term effects on pain, function, and mobility in non-specific low back pain. PeerJ. 2021 Mar 15;9:e10706. doi: 10.7717/peerj.10706. eCollection 2021. PMID 33777508
- [Background] Guo X, Li L, Yan Z, Li Y, Peng Z, Yang Y, Zhang Y, Schmitz C, Feng Z. Efficacy and safety of treating chronic nonspecific low back pain with radial extracorporeal shock wave therapy (rESWT), rESWT combined with celecoxib and eperisone (C + E) or C + E alone: a prospective, randomized trial. J Orthop Surg Res. 2021 Dec 4;16(1):705. doi: 10.1186/s13018-021-02848-x. PMID 34863239
- [Background] Shah SG, Kage V. Effect of Seven Sessions of Posterior-to-Anterior Spinal Mobilisation versus Prone Press-ups in Non-Specific Low Back Pain - Randomized Clinical Trial. J Clin Diagn Res. 2016 Mar;10(3):YC10-3. doi: 10.7860/JCDR/2016/15898.7485. Epub 2016 Mar 1. PMID 27134987
- [Background] Babina R, Mohanty PP, Pattnaik M. Effect of thoracic mobilization on respiratory parameters in chronic non-specific low back pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2016 Feb 19;29(3):587-95. doi: 10.3233/BMR-160679. PMID 26966825
- [Background] Riley SP, Tafuto V, Cote M, Brismee JM, Wright A, Cook C. Reliability and relationship of the fear-avoidance beliefs questionnaire with the shoulder pain and disability index and numeric pain rating scale in patients with shoulder pain. Physiother Theory Pract. 2019 May;35(5):464-470. doi: 10.1080/09593985.2018.1453004. Epub 2018 Mar 20. PMID 29558227